CLINICAL TRIAL: NCT00212979
Title: The Accurate Prediction of Renal Function in Kidney Transplant Recipients
Brief Title: Measuring Kidney Function in Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PSI Grant R03-59; REB Protocol #2003435-01H
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2009-02

CONDITIONS: Renal Transplant
Keywords: glomerular filtration rate; cystatin C; creatinine

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- non intervention study
  Interventions: Other: non intervention study

INTERVENTIONS:
Other: non intervention study

SUMMARY:
Kidney transplantation is the preferred treatment for permanent kidney failure. Following transplantation, the kidney function must be followed closely to detect problems so that investigations and appropriate treatment can be started early. Currently, function is monitored with the use of serum creatinine. In clinical trials involving kidney transplant recipients, markers of kidney function, such as serum creatinine, are increasingly being used as outcomes to evaluate new treatments. However, serum creatinine is not very accurate or sensitive at detecting change in kidney transplant function. Newer methods of evaluating kidney function, such as the Modification of Diet in Renal Disease (MDRD) equation and cystatin C, are known to be accurate markers of function in patients with non-transplant kidney disease. This study will compare the MDRD estimate and cystatin C estimate of kidney function with an accepted method (radioisotope clearance study) of measuring true kidney function in 250 renal transplant patients. Each patient will have 2 measurements made at least 3 months apart to determine the accuracy and responsiveness to change over time for the MDRD equation and cystatin C. If the results demonstrate that these new methods are accurate then clinical care and research studies involving transplant patients will be greatly enhanced. Patients and physicians would have a simple test that could detect problems earlier and more precisely monitor response to treatment leading to improved outcomes for renal transplant recipients.

DETAILED DESCRIPTION:
Background and Hypothesis:

Short-term outcomes in renal transplantation, such as the acute rejection rate, have improved dramatically over the past decade. Unfortunately, this success has made it more difficult to evaluate new therapies in kidney transplantation. Markers of kidney function, such as serum creatinine and creatinine clearance, are now being used to evaluate kidney transplant function. However, serum creatinine and creatinine clearance have many limitations and correlate poorly with the glomerular filtration rate (GFR). The Modification of Diet in Renal Disease (MDRD) formula has been shown to be very accurate at predicting GFR in patients with kidney disease who don't have renal transplants. Cystatin C, a novel marker of renal function, has also been shown to be accurate in transplant and non-transplant patients. However, the MDRD formula and cystatin C have not been properly validated in a large sample of renal transplant recipients.

Objectives:

The primary objective of this study is to determine if the MDRD formula accurately predicts GFR in renal transplant recipients. Secondary objectives of the study will determine whether: the MDRD formula is responsive to change in GFR over time, cystatin C accurately predicts GFR, or the MDRD formula is more accurate than other estimating equations in renal transplant recipients.

Research Plan:

A prospective cohort design will be used. Eligible adult renal transplant recipients at least 3 months post-transplantation will have serum creatinine, albumin, urea, cystatin C, 24-hour urine excretion of urea, 24-hour urine excretion of creatinine, 24-hour urine excretion of protein and GFR measured at study entry and at least 3 months later. GFR will be measured using 99Tc-DTPA. Estimates of the GFR will be made with the MDRD equation and other estimating equations. Renal function will also be assessed by measuring the urinary creatinine clearance and the combined urea and creatinine clearance. The primary analysis will determine the accuracy (proportion of GFR estimates that lie within 30% of measured GFR) of the MDRD equation. Secondary analyses will be performed to determine the bias (mean difference between the measured GFR and estimated GFR) and precision (standard deviation of the difference between the measured and estimated GFR) of the MDRD equation as well as the bias and precision of the change in GFR over twelve months. Similar analyses will be performed for cystatin C and other estimating equations.

Importance of Study:

New methods to accurately measure GFR are needed for both clinical care and research studies involving renal transplant recipients. As new therapies and immunosuppressive strategies become available, a simple and accurate means (such as the MDRD equation) to assess response to therapy will be invaluable. Markers of kidney function (serum creatinine, predicted GFR) are already being used in clinical trials involving renal transplant recipients without appropriate evaluation. The proper validation of equations to predict GFR in transplant recipients must be carried before they can be widely accepted in practice or for use in research protocols. If this study shows that the MDRD equation (or other marker of kidney function) is accurate in transplant patients then we can confidently move forward and use these validated measures of GFR in patient care and future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age.
* At least 6 months post-renal transplantation.

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Pregnant or breastfeeding
* Acute rejection within the preceding three months
* Likely to die from another comorbid disease within the next three months
* Likely to require dialysis or repeat transplantation within the next three months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg A Knoll, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada